CLINICAL TRIAL: NCT05650281
Title: Silent Progression Monitoring in Extreme Phenotypes. SP-MS, Despite an Effective Early Highly Active Treatment as a Paradigm SPAM Study (Silent Progression Activity Monitoring)
Brief Title: Silent Progression Activity Monitoring - SPAM Study
Acronym: SPAM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22Neuro03
Record Dates: First submitted 2022-08-08; First posted 2022-12-14 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with RRMS (2017 Mc Donald criteria) treated with highly active treatment in the first 5 years of symptoms onset, at least 1 year, with an EDSS below 4
  Interventions: Other: NO INTERVENTION

INTERVENTIONS:
Other: NO INTERVENTION — NO INTERVENTION

SUMMARY:
Real-World Data (RWD) exploring the natural history of MS suggested that relapses do not significantly influence the progression of irreversible disability. Disability progression independent of relapses activity (PIRA) has been confirmed as a frequent relapsing-remitting multiple sclerosis (RRMS) phenomenon based on Randomized Clinical Trials (RCT). Recently, RWD demonstrated that the absence of markers of inflammation (No Evidence of Disease Activity (NEDA) at 2 years did not predict long-term stability. Silent progression has been proposed to describe the insidious disability that accrues many patients who satisfy traditional criteria for relapsing-remitting MS. In this study, the investigators would like to evaluate the occurrence of the SPMS in a population of RRMS patient with an Highly Active Treatment (HAT).

ELIGIBILITY:
INCLUSION CRITERIA: - Patients with RRMS (2017 Mc Donald criteria) treated with highly active treatment in the first 5 years of symptoms onset, at least 1 year, with an EDSS below 4

* HAT start after April 12th 2007 (availability of Natalizumab)
* Naive or failure (or intolerability) to 1 or more first line DMT (injectables, teriflunomide, DMF).
* EDSS < or equal 4 when starting HAT EXCLUSION CRITERIA:
* Progressive relapsing MS at baseline
* Clinical or basic MRI data unavailable after on-site visit.
* MS diagnostic > 5 years at baseline
* Immunosuppressive drugs (Azathioprine, Cyclophosphamide, Mycophenolate, Methotrexate) prescribed before HAT initiation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with RRMS (2017 Mc Donald criteria) treated with highly active treatment in the first 5 years of symptoms onset, at least 1 year, with an EDSS below 4
Sampling Method: Non-Probability Sample
Enrollment: 2230 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Determination of baseline clinical markers associated with SPMS diagnosis despite an early, practical, Highly Active Treatment. | Baseline: beginning of highly active treatment
  Age in years
Determination of baseline clinical markers associated with SPMS diagnosis despite an early, practical, Highly Active Treatment. | Baseline: beginning of highly active treatment
  Disease duration (which should be <5 years) in months
Determination of baseline clinical markers associated with SPMS diagnosis despite an early, practical, Highly Active Treatment. | Baseline: beginning of highly active treatment
  Expanded Disability Status Scale (EDSS) (which must be <4)
Determination of baseline MRI markers associated with SPMS diagnosis despite an early, practical, Highly Active Treatment. | Baseline: beginning of highly active treatment
  new T2 lesion(s) on brain MRI and spinal cord MRI (if available)
Determination of baseline MRI markers associated with SPMS diagnosis despite an early, practical, Highly Active Treatment. | Baseline: beginning of highly active treatment
  gadolinium enhancement on brain MRI and spinal cord MRI (if available)
Determination of baseline clinical markers associated with SPMS diagnosis despite an early, practical, Highly Active Treatment. | Baseline: beginning of highly active treatment
  Interval time between the first and the second relapse in months
Determination of baseline clinical markers associated with SPMS diagnosis despite an early, practical, Highly Active Treatment. | Baseline: beginning of highly active treatment
  Reason for HAT: naive, or switch
Determination of baseline clinical markers associated with SPMS diagnosis despite an early, practical, Highly Active Treatment. | Baseline: beginning of highly active treatment
  Number of relapses since MS onset
Determination of baseline clinical markers associated with SPMS diagnosis despite an early, practical, Highly Active Treatment. | Baseline: beginning of highly active treatment
  DMT administered since MS onset: number of DMT and type
Determination of baseline MRI markers associated with SPMS diagnosis despite an early, practical, Highly Active Treatment. | Baseline: beginning of highly active treatment
  More than 9 T2 lesions on MRI
Determination of baseline MRI markers associated with SPMS diagnosis despite an early, practical, Highly Active Treatment. | Baseline: beginning of highly active treatment
  At least 1 periventicular T2 lesion on MRI
Determination of baseline MRI markers associated with SPMS diagnosis despite an early, practical, Highly Active Treatment. | Baseline: beginning of highly active treatment
  At least 3 periventicular T2 lesions on MRI
Determination of baseline MRI markers associated with SPMS diagnosis despite an early, practical, Highly Active Treatment. | Baseline: beginning of highly active treatment
  At least 1 infratentorial T2 lesion on MRI
Determination of baseline MRI markers associated with SPMS diagnosis despite an early, practical, Highly Active Treatment. | Baseline: beginning of highly active treatment
  At least 1 spinal cord T2 lesion on MRI
Determination of baseline MRI markers associated with SPMS diagnosis despite an early, practical, Highly Active Treatment. | Baseline: beginning of highly active treatment
  At least 1 gadolinium enhancement T1 lesion on MRI

SECONDARY OUTCOMES:
To determine re-baseline clinical markers associated with SPMS diagnosis despite an early, practical, HAT. | Re-baseline definition: any patient with at least an EDSS and MRI examination performed 12 months after HAT onset. +/- 6 months (from 6 to 18 months).
  Age in years
To determine re-baseline clinical markers associated with SPMS diagnosis despite an early, practical, HAT. | Re-baseline definition: any patient with at least an EDSS and MRI examination performed 12 months after HAT onset. +/- 6 months (from 6 to 18 months).
  Disease duration (which should be <5 years) in months
To determine re-baseline clinical markers associated with SPMS diagnosis despite an early, practical, HAT. | Re-baseline definition: any patient with at least an EDSS and MRI examination performed 12 months after HAT onset. +/- 6 months (from 6 to 18 months).
  EDSS (which must be <4) +/- 3 months
To determine re-baseline MRI markers associated with SPMS diagnosis despite an early, practical, HAT. | Re-baseline definition: any patient with at least an EDSS and MRI examination performed 12 months after HAT onset. +/- 6 months (from 6 to 18 months).
  new T2 lesion(s) on brain MRI and spinal cord MRI (if available)
To determine re-baseline MRI markers associated with SPMS diagnosis despite an early, practical, HAT. | Re-baseline definition: any patient with at least an EDSS and MRI examination performed 12 months after HAT onset. +/- 6 months (from 6 to 18 months).
  gadolinium enhancement on brain MRI and spinal cord MRI (if available)
To determine re-baseline MRI markers associated with SPMS diagnosis despite an early, practical, HAT. | Re-baseline definition: any patient with at least an EDSS and MRI examination performed 12 months after HAT onset. +/- 6 months (from 6 to 18 months).
  Interval time between the first and the second relapse in months
To determine re-baseline MRI markers associated with SPMS diagnosis despite an early, practical, HAT. | Re-baseline definition: any patient with at least an EDSS and MRI examination performed 12 months after HAT onset. +/- 6 months (from 6 to 18 months).
  Number of relapses since MS onset
To determine re-baseline MRI markers associated with SPMS diagnosis despite an early, practical, HAT. | Re-baseline definition: any patient with at least an EDSS and MRI examination performed 12 months after HAT onset. +/- 6 months (from 6 to 18 months).
  Number of relapse before baseline
To determine re-baseline MRI markers associated with SPMS diagnosis despite an early, practical, HAT. | Re-baseline definition: any patient with at least an EDSS and MRI examination performed 12 months after HAT onset. +/- 6 months (from 6 to 18 months).
  Disease Modifying Therapies (DMT) administered since MS onset
To determine re-baseline MRI markers associated with SPMS diagnosis despite an early, practical, HAT. | Re-baseline definition: any patient with at least an EDSS and MRI examination performed 12 months after HAT onset. +/- 6 months (from 6 to 18 months).
  More than 9 T2 lesions on MRI
To determine re-baseline MRI markers associated with SPMS diagnosis despite an early, practical, HAT. | Re-baseline definition: any patient with at least an EDSS and MRI examination performed 12 months after HAT onset. +/- 6 months (from 6 to 18 months).
  At least 1 periventicular T2 lesion on MRI
To determine re-baseline MRI markers associated with SPMS diagnosis despite an early, practical, HAT. | Re-baseline definition: any patient with at least an EDSS and MRI examination performed 12 months after HAT onset. +/- 6 months (from 6 to 18 months).
  At least 3 periventicular T2 lesion on MRI
To determine re-baseline MRI markers associated with SPMS diagnosis despite an early, practical, HAT. | Re-baseline definition: any patient with at least an EDSS and MRI examination performed 12 months after HAT onset. +/- 6 months (from 6 to 18 months).
  At least 1 infratentorial T2 lesion on MRI
To determine re-baseline MRI markers associated with SPMS diagnosis despite an early, practical, HAT. | Re-baseline definition: any patient with at least an EDSS and MRI examination performed 12 months after HAT onset. +/- 6 months (from 6 to 18 months).
  At least 1 spinal cord T2 lesion on MRI
To determine re-baseline clinical and MRI markers associated with SPMS diagnosis despite an early, practical, HAT. | Re-baseline definition: any patient with at least an EDSS and MRI examination performed 12 months after HAT onset. +/- 6 months (from 6 to 18 months).
  At least 1 gadolinium enhancement T1 lesion on MRI
Detremination of the impact of different definition of SPMS according to the clinician | Re-baseline definition: any patient with at least an EDSS and MRI examination performed 12 months after HAT onset. +/- 6 months (from 6 to 18 months).
  The definition of SPMS according to the clinician : neurological episode = start of progression as assessed by the time to develop SPMS in years.
Dertermination of the impact of different definition of SPMS according to Lublin. | at 5 years
  The definition of SPMS according to Lublin : progressive accumulation of disability after a primary relapsing course which must be confirmed at least 6 months after, as assessed by the time to develop SPMS in years.
Dertermination of the impact of different definition of SPMS according to Lorscheider. | at 5 years
  The definition of SPMS according to Lorscheider: with a minimum EDSS of 4 , an increase by 1 point if the EDSS was between 4 and 5.5, or an increase by 0.5 points if the EDSS was above 5.5, confirmed after 3 months., as assessed by the time to develop SPMS in years.
Analyze of the influence of NEDA (No Evidence of Disease activity) | at baseline and at 5 years
  The disease activity will be evalued by the NEDA score
Analyze of the influence of MEDA (Mild Evidence of Disease Activity) | at baseline and at 5 years
  The disease activity will be evalued by the MEDA score
To find a composite score usable at baseline when prescribing early HAT in clinical practice to predict early SPMS | at 5 years
  All baseline variables will be evaluated in association with the prescriptio of an early HAT to predict early SPMS.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No